CLINICAL TRIAL: NCT01783236
Title: A Double-blind, Randomized, Placebo-controlled Study to Compare the Effectiveness of IV Acetaminophen Administered Intra-operatively in Reducing the Use of Opiates to Treat Post-operative Pain
Brief Title: Analgesic Efficacy of Intravenous Acetaminophen After Video-assisted Thoracic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1204012295
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Lung Tumor
Keywords: VATS; thoracic surgery; acetaminophen; ofirmev; lung surgery; thoracoscopic; intravenous acetaminophen
MeSH Terms: conditions — Lung Neoplasms | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Placebo (Placebo Comparator): Subjects will receive a saline placebo infusion administered over 15 minutes every 6 hours for 24 hours.
  Interventions: Drug: Saline Placebo
- IV Acetaminophen (Active Comparator): Subjects will receive an infusion of 1 g of intravenous acetaminophen administered over 15 minutes every 6 hours for 24 hours with a maximum dose of 4 grams.
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — 1000mg IV Ofirmev given every six hours for a total of four doses.
  Other Names: Ofirmev; Paracetamol
  Arms: IV Acetaminophen
Drug: Saline Placebo — Normal saline placebo given every six hours for a total of four doses if randomized to the placebo arm.
  Other Names: Normal saline solution
  Arms: Saline Placebo

SUMMARY:
We will study the efficacy of FDA approved intravenous (IV) acetaminophen ("Ofirmev", © 2011 Cadence Pharmaceuticals, Inc.) in reducing opioid consumption after minimally invasive thoracic surgery in a double blind randomized trial. This drug has been shown in Europe to reduce the need for patient controlled analgesia and the total dose of opioids, which have serious side effects in thoracic surgery patients. We will compare the use of IV patient-controlled morphine (PCA) in two groups of subjects in treating postoperative pain. We will determine if IV acetaminophen reduces post-operative morphine requirements (primary end point). We will also assess subject pain scores and post-operative complications associated with pain management as secondary end points. Our hypothesis is that the study arm receiving intravenous acetaminophen will have lower total morphine consumptions compared to the placebo group.

DETAILED DESCRIPTION:
We will study the efficacy of FDA approved intravenous (IV) acetaminophen ("Ofirmev", © 2011 Cadence Pharmaceuticals, Inc.) in reducing opioid consumption after minimally invasive thoracic surgery in a double blind randomized trial. This drug has been shown in Europe to reduce the need for patient controlled analgesia and the total dose of opioids, which have serious side effects in thoracic surgery patients. We will compare the use of IV patient-controlled morphine (PCA) in two groups of subjects in treating postoperative pain. One group of subjects will receive IV acetaminophen every six hours beginning within 30 minutes before surgical end time and continuing for 24 hours plus IV morphine PCA, and the other group will receive IV placebo every six hours plus IV morphine PCA, a standard treatment for postoperative pain. We will determine if IV acetaminophen reduces post-operative morphine requirements (primary end point). We will also assess subject pain scores and post-operative complications associated with pain management as secondary end points. Our hypothesis is that the study arm receiving intravenous acetaminophen will have lower total morphine consumptions compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Any elective VATS patients with low probability of conversion to thoracotomy as determined by surgery.
* Ages 18-99
* American Society of Anesthesiologists Physical Status I-III, hemodynamically stable
* Male or female

Exclusion Criteria:

* Age less than 18.
* Patient refusal
* High probability of conversion to thoracotomy as determined by surgeon
* Conversion of procedure to thoracotomy (subjects will be withdrawn if VATS procedure is converted to thoracotomy, as thoracotomy is more invasive and will likely require additional analgesia such as neuraxial and regional anesthesia).
* Scheduled procedure of VATS Pleurodesis/decortication
* History of Interstitial Lung Disease
* Emergency case
* Known allergy/adverse reaction to acetaminophen, morphine, or fentanyl
* History of drug or alcohol abuse
* Patients on preoperative analgesic therapy within one week of surgery
* Contraindication to self administered morphine (unable to understand PCA)
* Need for postoperative mechanical ventilation
* Necessary major deviation for intraoperative study protocol as per the discretion of the intraoperative attending anesthesiologist
* History of congestive heart failure, renal failure, liver failure
* Pregnant or breastfeeding women
* Weight less than 51 kg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Hemmings, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- See also: Label information for acetaminophen (ofirmev) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/022450lbl.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline Placebo | IV Acetaminophen
Started | 8 | 8
Completed | 6 | 8
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Placebo | IV Acetaminophen | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (13.18) | 64.6 (8.23) | 61.8 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Morphine Consumption (mg)
Description: How much morphine the subject consumes in the first 24 hours after surgery (mg).
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Saline Placebo | IV Acetaminophen
Number analyzed (Participants) | 6 | 8
mg | 34.5 [21 to 98] | 44 [23 to 61.5]

2. Secondary Outcome: Total Number of PCA Requests in First 24 Hours Post-Operation
Description: The total number of Patient Controlled Analgesic (PCA) requests in the first 24 hours after the conclusion of the subject's operation
Time Frame: 24 hours post-operation
Measure: Median (Inter-Quartile Range); unit: PCA requests
Arm/Group | Saline Placebo | IV Acetaminophen
Number analyzed (Participants) | 6 | 8
PCA requests | 41 [17 to 144] | 43 [25 to 85]

3. Secondary Outcome: VAS Pain Score 2 Hours Post Operation
Description: 2 hours after the conclusion of their operation,participants were asked to draw a vertical line on the VAS to indicate their level of pain, which was then converted into millimeters for interpretations. Scores ranged from 0-100mm. VAS pain score identifies two extremes on a 10 centimeter horizontal line; the extremes are labeled "No Pain" (score of 0) and "Worst possible pain" (score of 100).
Time Frame: 2 Hours Post Operation
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Saline Placebo | IV Acetaminophen
Number analyzed (Participants) | 8 | 8
mm | 75.5 [59 to 87.5] | 49 [49 to 49]

4. Secondary Outcome: VAS Pain Score 6 Hours Post-Operation
Description: 6 hours after the conclusion of their operation, participants were asked to draw a vertical line on the VAS to indicate their level of pain, which was then converted into millimeters for interpretations. Scores ranged from 0-100mm. VAS pain score identifies two extremes on a 10 centimeter horizontal line; the extremes are labeled "No Pain" (score of 0) and "Worst possible pain" (score of 100).
Time Frame: 6 Hours Post-Operation
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Saline Placebo | IV Acetaminophen
Number analyzed (Participants) | 6 | 8
mm | 68.5 [65 to 71] | 39 [22.5 to 54.5]

5. Secondary Outcome: VAS Score 24 Hours Post-Operation
Description: 24 Hours after the conclusion of the subject's operation, participants were asked to draw a vertical line on the VAS to indicate their level of pain, which was then converted into millimeters for interpretations. Scores ranged from 0-100mm. VAS pain score identifies two extremes on a 10 centimeter horizontal line; the extremes are labeled "No Pain" (score of 0) and "Worst possible pain" (score of 100).
Time Frame: 24 hours post-operation
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Saline Placebo | IV Acetaminophen
Number analyzed (Participants) | 6 | 8
mm | 53 [29 to 67] | 16.5 [9 to 34.5]

ADVERSE EVENTS:
Time Frame: 24 hour study treatment period
Arm/Group | Saline Placebo | IV Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Placebo (N=8) | IV Acetaminophen (N=8)
Inadequate Pain Control (General disorders) | 2 (2) | 0 (0)
Lethargy (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No